CLINICAL TRIAL: NCT05388227
Title: Pole Walking Intervention Within Independent Living/Retirement Communities: Feasibility and Pilot
Brief Title: Pole Walking Intervention in Retirement Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Principal Investigator, Saija Kontulainen, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 141
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Fall Injury; Osteoporotic Fractures
Keywords: Patient-oriented; Exercise Intervention; Feasibility; Pilot
MeSH Terms: conditions — Osteoporotic Fractures | interventions — Nordic Walking

STUDY DESIGN:
Intervention Model Description: The feasibility phase of this study is a single-group trial with a primary purpose of assessing the feasibility of implementing a pole walking intervention within independent living/retirement communities. The pilot phase of this study is a two-arm, parallel-group, cluster-randomized, wait-list controlled trial with a primary purpose of assessing the efficacy of the pole walking intervention in improving physical activity, physical function, body composition, fear of falling, and health-related quality of life, and decreasing sedentary time in older adults living in independent living/retirement communities. In this phase, we anticipate enrolling 50 participants from residents of independent living/retirement communities. Communities will be randomly allocated to either the intervention or a wait-list control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pole walking intervention (Experimental): Will participate in supervised, group pole walking intervention sessions held at the participating communities, 2-3 times per week, for 20-60 minutes per session, over a 12-week period.
  Interventions: Other: Pole walking
- Wait-list control (No Intervention): Will continue life as usual during the 12-week period. However, after completing follow-up assessments, will also be offered the pole walking intervention at their communities.

INTERVENTIONS:
Other: Pole walking — The intervention will consist of group sessions held at the participating communities, 2-3 times per week, for 20-60 minutes per session, over a 12-week period. Pole walking exercises are tailored for participants and progressive in nature. Sessions will be led by trained peer, staff, or student instructors and conducted outdoors (indoors if weather conditions do not permit).
  Arms: Pole walking intervention

SUMMARY:
This patient-oriented, multi-site study aims to co-design and test a pole walking program with resident and staff representatives from participating independent living and retirement communities.

The first part of the study (feasibility phase) is a single-group trial designed to answer the main question: Is the pole walking program feasible in these settings? In this phase, all participants will take part in the program.

The second part of the study (pilot phase) is a two-group randomized trial that will assess whether the program helps improve physical activity, physical function, body composition, fear of falling, and health-related quality of life, while also reducing sedentary time (time spent sitting or being inactive) in older adults living in independent living and retirement communities. Communities will be randomly assigned to either start the program right away or join a wait-list control group.

The program will include supervised group sessions held at the participating communities, 2-3 times per week, for 20-60 minutes each session, over a 12-week period. Sessions will take place outdoors when possible, or indoors if the weather is not suitable.

After follow-up assessments are complete, participants in the control group will also be offered the pole walking program at their communities.

DETAILED DESCRIPTION:
Pole walking provides an attractive form of exercise therapy for older adults. It is a simple, well-tolerated, and effective means to improve overall functional fitness in older adults. Pole walking has improved upper and lower body muscle strength, cardiovascular endurance, and flexibility in community-dwelling older adults. It has been positively associated with balance, functional mobility, muscle strength, and aerobic exercise capacity in older adults. Pole walking is considered to offer a safe format for walking, as poles provide support and help with balance, and thus contribute to confidence in being active. However, there has not yet been a study assessing the feasibility and efficacy of a pole walking intervention in improving physical activity, physical function, body composition, fear of falling, and health-related quality of life, and decreasing sedentary time in older adults living in independent living/retirement communities.

This patient-oriented, multi-site study consists of a feasibility and a pilot phase. The feasibility phase is a single-arm trial that will assess the feasibility and safety of implementing a pole walking intervention within independent living/retirement communities. In this phase, all participants will receive the intervention. The pilot phase is a two-arm, parallel-group, cluster-randomized, wait-list controlled trial that will assess the efficacy of the pole walking intervention in improving physical activity, physical function, body composition, fear of falling, and health-related quality of life, and decreasing sedentary time in older adults living in independent living/retirement communities. In this phase, our target is to include 50 residents from independent living/retirement communities. Sites will be randomized to either the intervention or a wait-list control group. The intervention will consist of group sessions held at the participating communities, 2-3 times per week, for 20-60 minutes per session, over a 12-week period. Pole walking exercises are tailored for participants and progressive in nature. Sessions will be led by trained peer, staff, or student instructors and conducted outdoors (indoors if weather conditions do not permit). After completing follow-up assessments, participants in the control group will also be offered the pole walking program at their sites.

ELIGIBILITY:
Inclusion Criteria:

* Being an ambulatory resident in the independent living/retirement communities.
* Pass the Get Active Questionnaire. If the participant has heart conditions, angina during daily living, balance, and bone or joint problems, then a Physician Clearance Form is required to be filled out and signed by the participant's family physician.

Exclusion Criteria:

* Using assistive devices for mobility.
* Being active (moderate-to-vigorous physical activity ≥150 min/week).
* Diagnosed with Parkinson's disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of pole walking intervention - consent rate | After the completion of the study's feasibility phase (1 year)
  Assessed by calculating consent rate (%) as the percentage of participants assessed for eligibility who consented.
Feasibility of pole walking intervention - recruitment rate | After the completion of the study's feasibility phase (1 year)
  Assessed by calculating recruitment rate (participant/site/month) as the number of potentially eligible participants who consented divided by the number of recruiting sites and then divided by the number of months spent on recruitment.
Feasibility of pole walking intervention - retention rate | After the completion of the study's feasibility phase (1 year)
  Assessed by calculating retention rate (%) as the percentage of eligible participants enrolled in the study who received the allocated intervention and completed both baseline and follow-up assessments.
Feasibility of pole walking intervention - attendance rate | After the completion of the study's feasibility phase (1 year)
  Assessed by calculating attendance rate (%) as the percentage of available intervention sessions attended by each participant.
Feasibility of pole walking intervention - intervention acceptability score | Follow-up assessment sessions (after the 12-week intervention of the study's feasibility phase)
  Assessed by calculating intervention acceptability score (ranging from 1-5, with higher scores indicating greater acceptability of an intervention ) using the 4-item intervention acceptability measure.
Feasibility of pole walking intervention - intervention appropriateness score | Follow-up assessment sessions (after the 12-week intervention of the study's feasibility phase)
  Assessed by calculating intervention appropriateness score (ranging from 1-5, with higher scores indicating greater appropriateness of an intervention ) using the 4-item intervention appropriateness measure.
Feasibility of pole walking intervention - intervention feasibility score | Follow-up assessment sessions (after the 12-week intervention of the study's feasibility phase)
  Assessed by calculating intervention feasibility score (ranging from 1-5, with higher scores indicating greater feasibility of an intervention ) using the 4-item intervention feasibility measure.
Physical function - functional balance/mobility | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the timed "up & go" test.
Physical function - lower-body strength | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the 30-s chair stand test.
Health-related quality of life | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the 36-item short form survey, which provides a score ranging from 0-100 for each of its 8 scales (the higher the scale scores, the more favorable the corresponding health states).

SECONDARY OUTCOMES:
Safety of pole walking intervention | Follow-up assessment sessions (after the 12-week intervention of the study's feasibility phase)
  Assessed by the seriousness and relatedness to the intervention of recorded adverse events.
Physical function - functional capacity | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the 6-min walk test.
Physical function - upper-body strength | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the grip strength test.
Physical activity/sedentary time | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by 7-day accelerometry.
Fear of falling | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the 10-item falls efficacy scale, which provides a total score ranging from 10-100, with higher scores suggesting greater fear of falling.
Body composition - musculoskeletal properties of the lower leg | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the peripheral quantitative computed tomography.
Body composition - musculoskeletal properties of the forearm | Baseline and follow-up assessment sessions (before and after the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the peripheral quantitative computed tomography.

OTHER OUTCOMES:
Body composition - areal bone mineral density at the hip | Baseline assessment sessions (before the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the dual-energy X-ray absorptiometry.
Body composition - areal bone mineral density at the lumbar spine | Baseline assessment sessions (before the 12-week intervention of the study's feasibility and pilot phases)
  Assessed by the dual-energy X-ray absorptiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Saija A Kontulainen, PhD, Principal Investigator — Professor, College of Kinesiology, University of Saskatchewan
Locations (1):
- Saija Kontulainen, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No